CLINICAL TRIAL: NCT02061891
Title: Entire Danish Initiative To ImrpOve Revascularization Strategies (EDITORS) - A Randomised Evaluation of Clinical Outcome After Acute or Deferred Invasive Intervention Integrated With MDCT Imaging in Patients With Acute Coronary Syndromes
Brief Title: Very Early veRsus Deferred Invasive Evaluation Using Computerized Tomography in Patients With Acute Coronary Syndromes
Acronym: VERDICT-EDI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Klaus Fuglsang Kofoed, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2010-039; EDITORS (Other: The Danish Council for Strategic Research (09-066994))
Record Dates: First submitted 2014-02-06; First posted 2014-02-13 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Stenosis; Coronary Artery Disease; Acute coronary syndrome; Percutaneous Coronary Intervention; Multidetector Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferred invasive evaluation (Active Comparator): Deferred invasive coronary evaluation and revascularization (PCI/CABG) within 72 hours from time of clinical diagnosis (CONTROL group)
  Interventions: Procedure: Invasive coronary evaluation (Deferred)
- Very early invasive evaluation (Experimental): Acute invasive coronary evaluation within 12 hours from time of diagnosis - INTERVENTION group
  Interventions: Procedure: Invasive coronary evaluation (Acute)

INTERVENTIONS:
Procedure: Invasive coronary evaluation (Deferred) — Invasive coronary angiography and revascularization (PCI/CABG)
  Arms: Deferred invasive evaluation
Procedure: Invasive coronary evaluation (Acute) — Invasive coronary angiography and revascularization (PCI/CABG)
  Arms: Very early invasive evaluation

SUMMARY:
The aim of this study is to evaluate if acute invasive coronary evaluation and treatment conducted within 12 hours of diagnosis improves clinical outcome compared to a deferred, subacute strategy in patients with unstable angina pectoris (UAP) / non-ST segment elevation myocardial infarction (NSTEMI) Acute coronary syndrome (ACS) Furthermore, in an observational design the potential clinical benefit of coronary computed tomography angiography (CCTA) to select patients for invasive investigation and treatment in the two treatment arms (acute vs deferred) is evaluated.

The following main hypothesis will be tested:

* Very early invasive coronary investigation improves clinical outcome in patients with UAP/NSTEMI-ACS
* CCTA performed before invasive coronary investigation will improve clinical management of patients with UAP/NSTEMI-ACS

DETAILED DESCRIPTION:
MATERIAL Consecutive patients suspected of UAP/NSTEMI will be screened for participation in the study. Only patients deemed clinically suited for invasive coronary evaluation and treatment will be included. A total of 2500 patients will be included in the trial at Departments of Cardiology of Danish Hospitals.

METHODS If the patients accept participation in the trial a computerized 1:1 randomization for acute invasive coronary evaluation (Intervention group - within 12 hours from time of diagnosis) or for deferred invasive evaluation (Control group - no later than 72 hours from time of diagnosis). All included patients undergo CCTA prior to invasive coronary evaluation, except for patient with moderately reduced renal function (se below). The treating invasive cardiologist will remain blinded to observational CCTA data. Patients with endstage renal disease in dialysis may undergo CCTA. CCTA data recorded as part of the research protocol will not be made available for the treating physician.

SECONDARY EXCLUSION Based on post-hoc expert clinical evaluation patients not having UAP/NSTEMI-ACS (arrythmias, pulmonary oedema, missed STEMI, pneumonia, Pulmonary emboli) will be excluded from analysis of difference between outcome measures in treatment strategy groups.

STATISTICAL METHODS Patients with UAP/NSTEMI-ACS are based on previous studies expected to have an event rate of 15% within 1 year and 50% at 4 years of the primary combined endpoint: all cause mortality, non-fatal recurrent myocardial infarction, hospitalisation for refractory ischemia or heart failure. In order to demonstrate a reduction of 25% within 3 years 711 patients in each group are needed. The study is powered to detect a clinical relevant reduction in mortality or heart failure hospitalization with a total of 2500 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical suspicion of of UAP/NSTEMI acute coronary syndrome deemed suitable for invasive evaluation and treatment will be included in the study.

* Age> 18 years
* At least one of the following:
* ECG abnormalities suggestive of myocardial ischemia (newly developed ST segment depression, horizontal or descending >= 0,05mV in two anatomically adjacent leads and/or T-wave inversion >0,01 mV in two leads with prominent R wave or R/S ratio >1
* Elevated myocardial ischemia biomarkers (Troponin, CK-MB)

Exclusion Criteria:

* Pregnancy
* Circumstances preventing the patient from reading and/or understanding the research protocol information
* Clinical indication for acute invasive coronary angiography - severe chest pain despite intravenous nitroglycerin infusion or hemodynamic instability
* Expected survival of less than 1 year
* Known allergy/hypersensitivity of pharmacological platelet inhibitors and/or iodine contrast that cannot be prevented medically

Patients with known eGFR below 60 ml/min will not undergo CCTA, whereas patients in dialysis will undergo the entire study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-06 (Actual); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Composite clinical endpoint | 3 years
  Composite endpoint of all cause mortality, non-fatal recurrent acute myocardial infarction, hospitalisation for refractory ischemia (acute coronary syndrome) or heart failure

SECONDARY OUTCOMES:
Bleeding | During index hospitalization - an expected average of 5 days
  Major and minor bleeding according to TIMI and BARC classification systems
Non-bleeding, invasive procedure related complications | During index hospitalization - an expected average of 5 days
  Invasive procedure related acute myocardial infarction, embolic stroke, cardiac arrest
Death | 3 and 5 years
  All-cause death
Non-fatal acute myocardial infarction | 3 and 5 years
Hospital admittance due to refractory myocardial ischemia (acute coronary syndrome) | 3 and 5 years
Repeat coronary revascularization | 3 and 5 years
  Recorded from 30 days post-index procedure
Hospital admittance due to left ventricular heart failure | 3 and 5 years
GRACE Risk Score | 3 and 5 years
  All primary and secondary endpoints stratified by GRACE score at a threshold of 140

OTHER OUTCOMES:
CCTA diagnostic accuracy | Within 30 days after performed CCTA and ICA
  Determinants of diagnostic accuracy of CCTA for the identification of >50% and >70% coronary artery stenosis by invasive coronary angiography in both treatment strategy groups
CCTA guided treatment strategy | Within 30 days after performed CCTA and ICA
  Prediction of clinical treatment strategy based on CCTA - and the potential value of CCTA guided triage in terms of optimized patient management. Evaluation will be performed blinded to ICA findings.
CCTA prediction of clinical outcome | 3 and 5 years
  Clinical prognostic value of coronary pathology, cardiac and non-cardiac pathology identified by CCTA

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Køber, MD, DmSc, Study Chair — Department of Cardiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Denmark
Locations (1):
- Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Navarese EP, Gurbel PA, Andreotti F, Tantry U, Jeong YH, Kozinski M, Engstrom T, Di Pasquale G, Kochman W, Ardissino D, Kedhi E, Stone GW, Kubica J. Optimal timing of coronary invasive strategy in non-ST-segment elevation acute coronary syndromes: a systematic review and meta-analysis. Ann Intern Med. 2013 Feb 19;158(4):261-70. doi: 10.7326/0003-4819-158-4-201302190-00006. PMID 23420234
- [Background] Mehta SR, Granger CB, Boden WE, Steg PG, Bassand JP, Faxon DP, Afzal R, Chrolavicius S, Jolly SS, Widimsky P, Avezum A, Rupprecht HJ, Zhu J, Col J, Natarajan MK, Horsman C, Fox KA, Yusuf S; TIMACS Investigators. Early versus delayed invasive intervention in acute coronary syndromes. N Engl J Med. 2009 May 21;360(21):2165-75. doi: 10.1056/NEJMoa0807986. PMID 19458363
- [Background] Kristensen TS, Kofoed KF, Kuhl JT, Nielsen WB, Nielsen MB, Kelbaek H. Prognostic implications of nonobstructive coronary plaques in patients with non-ST-segment elevation myocardial infarction: a multidetector computed tomography study. J Am Coll Cardiol. 2011 Jul 26;58(5):502-9. doi: 10.1016/j.jacc.2011.01.058. PMID 21777748
- [Derived] Ratcovich H, Sadjadieh G, Linde JJ, Joshi FR, Kelbaek H, Kofoed KF, Kober L, Hansen PR, Torp-Pedersen C, Elming H, Gislason GH, Hofsten DE, Engstrom T, Holmvang L. Coronary CT and timing of invasive coronary angiography in patients >/=75 years old with non-ST segment elevation acute coronary syndromes. Heart. 2023 Feb 23;109(6):457-463. doi: 10.1136/heartjnl-2022-321640. PMID 36351794
- [Derived] Butt JH, Kofoed KF, Kelbaek H, Hansen PR, Torp-Pedersen C, Hofsten D, Holmvang L, Pedersen F, Bang LE, Sigvardsen PE, Clemmensen P, Linde JJ, Heitmann M, Hove JD, Abdulla J, Gislason G, Engstrom T, Kober L. Importance of Risk Assessment in Timing of Invasive Coronary Evaluation and Treatment of Patients With Non-ST-Segment-Elevation Acute Coronary Syndrome: Insights From the VERDICT Trial. J Am Heart Assoc. 2021 Oct 5;10(19):e022333. doi: 10.1161/JAHA.121.022333. Epub 2021 Sep 29. PMID 34585591
- [Derived] Kofoed KF, Engstrom T, Sigvardsen PE, Linde JJ, Torp-Pedersen C, de Knegt M, Hansen PR, Fritz-Hansen T, Bech J, Heitmann M, Nielsen OW, Hofsten D, Kuhl JT, Raymond IE, Kristiansen OP, Svendsen IH, Dominguez Vall-Lamora MH, Kragelund C, Hove JD, Jorgensen T, Fornitz GG, Steffensen R, Jurlander B, Abdulla J, Lyngbaek S, Elming H, Therkelsen SK, Jorgensen E, Klovgaard L, Bang LE, Helqvist S, Galatius S, Pedersen F, Abildgaard U, Clemmensen P, Saunamaki K, Holmvang L, Gislason G, Kelbaek H, Kober LV. Prognostic Value of Coronary CT Angiography in Patients With Non-ST-Segment Elevation Acute Coronary Syndromes. J Am Coll Cardiol. 2021 Mar 2;77(8):1044-1052. doi: 10.1016/j.jacc.2020.12.037. PMID 33632478
- [Derived] Linde JJ, Kelbaek H, Hansen TF, Sigvardsen PE, Torp-Pedersen C, Bech J, Heitmann M, Nielsen OW, Hofsten D, Kuhl JT, Raymond IE, Kristiansen OP, Svendsen IH, Vall-Lamora MHD, Kragelund C, de Knegt M, Hove JD, Jorgensen T, Fornitz GG, Steffensen R, Jurlander B, Abdulla J, Lyngbaek S, Elming H, Therkelsen SK, Jorgensen E, Klovgaard L, Bang LE, Hansen PR, Helqvist S, Galatius S, Pedersen F, Abildgaard U, Clemmensen P, Saunamaki K, Holmvang L, Engstrom T, Gislason G, Kober LV, Kofoed KF. Coronary CT Angiography in Patients With Non-ST-Segment Elevation Acute Coronary Syndrome. J Am Coll Cardiol. 2020 Feb 11;75(5):453-463. doi: 10.1016/j.jacc.2019.12.012. PMID 32029126
- [Derived] Kofoed KF, Kelbaek H, Hansen PR, Torp-Pedersen C, Hofsten D, Klovgaard L, Holmvang L, Helqvist S, Jorgensen E, Galatius S, Pedersen F, Bang L, Saunamaki K, Clemmensen P, Linde JJ, Heitmann M, Wendelboe Nielsen O, Raymond IE, Kristiansen OP, Svendsen IH, Bech J, Dominguez Vall-Lamora MH, Kragelund C, Hansen TF, Dahlgaard Hove J, Jorgensen T, Fornitz GG, Steffensen R, Jurlander B, Abdulla J, Lyngbaek S, Elming H, Therkelsen SK, Abildgaard U, Jensen JS, Gislason G, Kober LV, Engstrom T. Early Versus Standard Care Invasive Examination and Treatment of Patients With Non-ST-Segment Elevation Acute Coronary Syndrome. Circulation. 2018 Dec 11;138(24):2741-2750. doi: 10.1161/CIRCULATIONAHA.118.037152. PMID 30565996